CLINICAL TRIAL: NCT03521544
Title: Self-Myofascial Release in the Posterior Myofascial Chain in Healthy Subjects With a Foam Roller
Brief Title: Self-Myofascial Release in the Posterior Myofascial Chain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Director, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P1/01
Record Dates: First submitted 2018-04-12; First posted 2018-05-11 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Fasciae (Anatomy)--Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Plantar Fascia (Experimental): Self-myofascial release in the plantar fascia.
  Interventions: Other: Self-myofascial release
- Tricep surae fascia (Experimental): Self-myofascial release in the triceps surae fascia.
  Interventions: Other: Self-myofascial release
- Hamstrings fascia (Experimental): Self-myofascial release in the hamstrings fascia.
  Interventions: Other: Self-myofascial release
- Spine erectors and lumbar fascia (Experimental): Self-myofascial release in the spine erectors and lumbar fascia.
  Interventions: Other: Self-myofascial release
- Occipital and suboccipital fascia (Experimental): Self-myofascial release in the occipital and suboccipital fascia.
  Interventions: Other: Self-myofascial release
- Control group (No Intervention): Lay on a stretcher.

INTERVENTIONS:
Other: Self-myofascial release — The subjects roll a foam roller under a determinated part of the body to self-massage that area.
  Other Names: Foam rolling
  Arms: Hamstrings fascia; Occipital and suboccipital fascia; Plantar Fascia; Spine erectors and lumbar fascia; Tricep surae fascia

SUMMARY:
The study investigates the relation between different segments of the posterior myofascial chain of the human body.

The intervention consists on apply self-myofascial release with a foam roller in one of the segments of the posterior myofascial chain of the participants, and then see if the treatment has produced any changes in the hamstrings, gastrocnemius and soleus flexibility.

DETAILED DESCRIPTION:
The study investigates the relation between different segments of the posterior myofascial chain of the human body.

The intervention consists on apply self-myofascial release with a foam roller in one of the segments of the posterior myofascial chain, and then see if the treatment has produced any changes in the hamstrings, gastrocnemius and soleus flexibility.

ELIGIBILITY:
Exclusion Criteria:

* Pregnant women
* Musculoskeletal problems in the last month
* Surgical interventions in he knee, hip, ankle, back or neck in tha last 6 months
* Psychological or nervous alterations
* Uncomprehension of the study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Hamstrings flexibility change | 0 seconds, 30 seconds, 2 minutes, 5 minutes, 10 minutes
  Measurement of the hamstrings flexibility change through Sit and Reach Test

SECONDARY OUTCOMES:
Triceps surae flexibility change | 0 seconds, 10 minutes
  Measurement of the triceps surae flexibility change using the Lunge Test.
Fatigue | 10 minutes
  Fatigue subjective sensation using the Modified Borg Scale

CONTACTS AND LOCATIONS:
Overall Officials: Albert Pérez Bellmunt, PhD, Principal Investigator — Anatomy lecturer
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided